CLINICAL TRIAL: NCT05941494
Title: Cerebral Hemodynamic and Metabolic Responses to Anesthesia and Vasopressors in Adult Surgery: A 2x2 Factorial Design Randomized Controlled Trial With Light-based Neuromonitoring (CHEM-FACT Study)
Brief Title: Cerebral Flow-metabolism Coupling During Adult Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jason Chui (Other)
Responsible Party: Sponsor-Investigator, Jason Chui, Anesthesiologist, Associate Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: CHEM FACT
Record Dates: First submitted 2023-07-04; First posted 2023-07-12 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Anesthesia
Keywords: Anesthesia Drugs; Vasopressors; Neuromonitoring
MeSH Terms: interventions — Propofol; Sevoflurane; Ephedrine; Phenylephrine

STUDY DESIGN:
Intervention Model Description: This is a prospective, 2x2 factorial design, blinded, randomized controlled study. Written informed consent will be obtained from all participants. We will recruit 80 adult patients (age >18 years old), who are ASA I-III and are scheduled for surgery under general anesthesia. We will randomize these patients into one of the four groups in 1:1:1:1 ratio for one of two choices of anesthetic maintenance agents and vasopressors.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcomes assessors will be blinded to the combination of anesthetic maintenance agents (propofol or sevoflurane) and vasopressors (phenylephrine or ephedrine) that were used during surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Propofol-based anesthetic maintenance with phenylephrine used as the vasopressor (Experimental): Propofol-based anesthetic maintenance with phenylephrine used as the vasopressor. Patient will receive propofol as their maintenance agent during surgery. The typical dose is 150-200 mg/kg/min. Patient will receive phenylephrine infusion as the primary vasopressor of choice. The typical dose of phenylephrine infusion is 10-40 mcg/min (dilution 100 mcg/ml).
  Interventions: Drug: Propofol; Drug: Phenylephrine
- Propofol-based anesthetic maintenance with ephedrine used as the vasopressor (Experimental): Propofol-based anesthetic maintenance with ephedrine used as the vasopressor. Patient will receive propofol as their maintenance agent during surgery. The typical dose is 150-200 mg/kg/min. The patient will receive ephedrine infusion as the primary vasopressor of choice. The typical dose of ephedrine infusion is 10-50 mg/hr (dilution 2 mg/ml).
  Interventions: Drug: Propofol; Drug: Ephedrine
- Sevoflurane-based anesthetic maintenance with phenylephrine used as the vasopressor (Experimental): Sevoflurane-based anesthetic maintenance with phenylephrine used as the vasopressor.
  Patient's anesthesia will be maintained with 1 MAC of sevoflurane during surgery. Patient will receive phenylephrine infusion as the primary vasopressor of choice. The typical dose of phenylephrine infusion is 10-40 mcg/min (dilution 100 mcg/ml).
  Interventions: Drug: Sevoflurane; Drug: Phenylephrine
- Sevoflurane-based anesthetic maintenance with ephedrine used as the vasopressor (Experimental): Sevoflurane-based anesthetic maintenance with ephedrine used as the vasopressor. Patient's anesthesia will be maintained with 1 MAC of sevoflurane during surgery. The patient will receive ephedrine infusion as the primary vasopressor of choice. The typical dose of ephedrine infusion is 10-50 mg/hr (dilution 2 mg/ml).
  Interventions: Drug: Sevoflurane; Drug: Ephedrine

INTERVENTIONS:
Drug: Propofol — Patient will receive propofol as their maintenance agent during surgery. The typical dose is 150-200 mg/kg/min.
  Other Names: Propofol for anesthesia maintenance
  Arms: Propofol-based anesthetic maintenance with ephedrine used as the vasopressor; Propofol-based anesthetic maintenance with phenylephrine used as the vasopressor
Drug: Sevoflurane — Patient's anesthesia will be maintained with 1 MAC of sevoflurane during surgery.
  Other Names: Sevoflurane for anesthesia maintenance
  Arms: Sevoflurane-based anesthetic maintenance with ephedrine used as the vasopressor; Sevoflurane-based anesthetic maintenance with phenylephrine used as the vasopressor
Drug: Ephedrine — The patient will receive ephedrine infusion as the primary vasopressor of choice. The typical dose of ephedrine infusion is 10-50 mg/hr (dilution 2 mg/ml).
  Other Names: Ephedrine as a vasopressor
  Arms: Propofol-based anesthetic maintenance with ephedrine used as the vasopressor; Sevoflurane-based anesthetic maintenance with ephedrine used as the vasopressor
Drug: Phenylephrine — Patient will receive phenylephrine infusion as the primary vasopressor of choice. The typical dose of phenylephrine infusion is 10-40 mcg/min (dilution 100 mcg/ml).
  Other Names: Phenylephrine as a vasopressor
  Arms: Propofol-based anesthetic maintenance with phenylephrine used as the vasopressor; Sevoflurane-based anesthetic maintenance with phenylephrine used as the vasopressor

SUMMARY:
The brain is a highly active organ that requires a large blood flow to function properly. Normally, blood flow is tightly linked to the brain's energy demands. However, during surgery, anesthesia can affect this relationship in different ways. Some types of anesthesia can decrease blood flow to the brain, while others can increase it. Anesthesiologists need to be careful to maintain adequate blood flow to the brain during surgery, especially when blood pressure drops. Drugs may be used to increase blood pressure, but some of these drugs can also affect blood flow to the brain. It is still unclear how to best maintain blood flow to the brain during surgery and how different types of anesthesia and drugs affect this process.

The study aims to assess the clinical utility of a new technique that uses light-based neuromonitoring to measure changes in cerebral blood flow and metabolism. The investigators will recruit 80 adult patients undergoing surgery under general anesthesia and randomize them into one of four groups to evaluate the effects of different anesthetic agents and vasopressors on brain hemodynamics and metabolism. The study will include patients over 18 years of age with no history of neurological conditions, substance abuse, or contraindications to cerebral oximetry devices or specific anesthetic agents. The patients will receive standard anesthesia care and be monitored with our light-based neuromonitoring system. This study aims to demonstrate the device's ability to detect changes in cerebral hemodynamic parameters related to anesthesia induction and systemic hypotension. This study will also evaluate the effects of anesthetic maintenance agents and vasopressors on cerebral hemodynamics and neurovascular coupling.

DETAILED DESCRIPTION:
The brain is a highly metabolic active organ, which receives approximately 15% of cardiac output with a normal cerebral blood ﬂow (CBF) of approximately 50 mL/100 g/min. In normal circumstances, CBF is tightly coupled to local cerebral metabolism. An increase of cerebral metabolic activity of one region of the brain will trigger a corresponding increase of blood ﬂow to that brain region. Conversely, a reduction of cerebral metabolic activity will lead to a reduction in blood ﬂow. This tightly controlled physiological phenomenon is known as ﬂow-metabolism coupling.

Flow-metabolism coupling is thought to be a feed-forward physiological protective mechanism wherein neuronal activity directly increases CBF, thereby matching the increased energy supply. In the event of cerebral hypoperfusion (i.e. reduction in CBF), brain vessels would be dilated in compensation and the local oxygen extraction fraction (OEF) would be increased. If cerebral hypoperfusion persists and is below the threshold, the activity of the brain cells would be suppressed, thereby resulting in the reduction of the cerebral metabolic rate (CMR) and cerebral metabolic requirement of oxygen (CMRO2). This flow-metabolism coupling mechanism is well studied using a PET scan in both healthy volunteers and patients with pathological conditions. Importantly, this physiological property of flow-metabolism in response to brain ischemia may be used as an earlier indicator of cerebral ischemia during surgery. In other words, monitoring that indicates a sudden drop in CMRO2 or increase in OEF may serve as an early marker of brain ischemia. However, due to technical limitations, bedside detection of such subtle physiological changes is challenging, especially in the intraoperative settings. In addition, many physiological, pathological, and pharmacological factors may affect this flow-metabolism coupling relationship and hence affect the interpretation of CMRO2/OEF changes as an indicator of brain ischemia. Additional studies are required to address how anesthetics may confound the interpretation.

Different anesthetic agents may alter flow-metabolism coupling in different ways. Cerebral metabolic rate is determined by a number of factors, including the functional state of the nervous system, anesthetic drugs and body temperature. The effect of individual anesthetic drugs on the CMR has been well studied. In short, most anesthetic drugs suppress the CMR in a dose-dependent manner, with the exception of ketamine and nitrous oxide (N2O). The anesthetic suppression of the CMR is mainly driven by the reduction of electrophysiologic activities. Previous studies have showed several anesthetics, including barbiturates, isoﬂurane, sevoﬂurane, desﬂurane, propofol, and etomidate can increase plasma concentrations and cause progressive suppression of EEG activity and a concomitant reduction in the CMR.

To further complicate the issue, during surgery, the anesthesiologist is required to maintain adequate cerebral perfusion pressure to ensure that there is sufficient CBF to meet metabolic demands. Induction of general anesthesia is often associated with a reduction in the mean arterial blood pressure(MAP) and cerebral perfusion pressure which is attributable to a decrease in cardiac output (CO) and systemic vascular resistance (SVR). Many intraoperative conditions such as blood loss and surgical positioning, may further compromise patient blood pressure and hence, CBF. Phenylephrine and ephedrine are commonly administered during neurosurgical procedures to counteract cardiovascular depression and treat anesthesia-related hypotension. Near-infrared spectroscopy (NIRS) studies in anesthetized patients suggest that phenylephrine reduces regional cerebral oxygen saturation (StO2) compared with ephedrine, despite a marked increase in the MAP. The results of these studies are conflicting and are various limitations.

NIRS has long been recognized as a promising neuromonitor due to the relative transparency of tissue to light in the near-infrared range and the dependency of light absorption on the oxygenation of haemoglobin, which provides a non-invasive method of measuring StO2. In addition, NIRS is extremely safe, inexpensive and provides real-time monitoring. Commercial systems are available and have been used for neuromonitoring during a variety of surgical procedures with an associated risk of brain injury, including coronary artery bypass and carotid endarterectomy.1,2 Despite the advantages of NIRS, its diagnostic accuracy for detecting intra-operative ischemia is controversial.3 A recent systematic review concluded that:

"NIRS has low sensitivity and high specificity to identify intra-operative ischaemia … Extracranial signal contribution was highly variable." 4

This conclusion reflects the two main limitations with commercial NIRS systems. First, the relationship between StO2 and ischemia is not direct since StO2 not only depends on CBF but also on the metabolic demand of the tissue. Second, light absorption in the scalp and skull is a major source of signal contamination. In fact, more than 80% of the NIRS signal originates from the extra-cerebral tissues since the distance from the skin surface to the brain ranges between 1.0 to 1.5 cm. As a result, hemodynamic changes in the superficial tissues can overshadow brain-related signals. Because of these two limitations, a specific StO2 threshold to identify intra-operative ischemia has not been established.

Our team has been developing technologies to tackle the two main limitations with commercial NIRS systems. With regards to enhancing depth sensitivity, the investigators have developed a time-resolved (tr)NIRS system that measures the time photons take to travel through tissue.5 Based on the principle that time equals distance, light that interrogates scalp and skull is recorded earlier than light that reaches the brain.

To provide continuous blood flow monitoring, the investigators have combined trNIRS with a complementary optical technology known as diffuse correlation spectroscopy (DCS). Instead of measuring light absorption, DCS measures temporal signal fluctuations caused by the movement of light scatterers, which in tissue is dominated by microvasculature blood flow (i.e. tissue perfusion).8 Like NIRS, DCS can be affected by signal changes in superficial tissue, although it has the intrinsic advantage that blood flow is considerably higher in the brain compared to the scalp (~ 5:1).9 To separate the two signal contributions, our system acquires data at two source-detector distances: a short distance to monitor scalp blood flow and a longer distance with greater sensitivity to CBF.10 The investigators have previously used DCS to monitor CBF stability in preterm infants during the first days of life and during cardiac surgery.11,12 A recent paper investigating the use of DCS to monitor CBF during carotid endarterectomy reported an average reduction in perfusion of 57% with clamping13.

Our hybrid trNIRS/DCS, which is shown has the ability to measure CBF and StO2 simultaneously. With this combination, oxygen metabolism in the brain, which is referred to as the cerebral metabolic rate of oxygen consumption (CMRO2), can be calculated by combining the two measurements.

Based on this new developed bed-side technique, the investigators plan to assess how CBF and CMRO2 change under general anesthesia and their responses toward phenylephrine and ephedrine during hypotension.

All study participants will be recruited and consented adhering to the local ethics guidelines. The attending anesthesiologists and the surgeons will not be blinded because of the nature of the intervention. However, patients and outcomes assessors will be blinded as to the treatment intervention. All patients will receive standard anesthesia care and the surgical and anesthetic management of the patients will be conducted in a standard fashion and will not be altered in this study. Anesthesia will be induced with fentanyl of 1-2 mcg/kg, propofol of 1.5-3 mg/kg, rocuronium of 0.6-0.9 mg/kg. Automatic blood pressure, electrocardiography, pulse oximetry, capnography, oesophageal temperature, and inspired and expired oxygen and CO2 concentration will be monitored. Controlled ventilation with 50% oxygen in air will be applied and the end-tidal CO2 levels will be maintained at 35-40 mmHg. The oxygen saturation is maintained above 96%. FiO2 can be increased if arterial desaturation occurs. Body temperature will be maintained above 36 ℃. After surgery, the patients will be extubated and transferred to the PACU. The depth of anesthesia will be continuously monitored either by bispectral index (BSI) or patient state index (PSI).

All patients will be monitored by the trNIRS/DCS device from anesthesia induction to completion of surgery. The NIRS sensor will be placed on the patient's forehead.

Before anesthesia induction, preoperative baseline cerebral hemodynamic and metabolic parameters such as ScO2, CBF, CMRO2, OEF will be measured for 1 minute. Monitoring will be continued during anesthesia induction and tracheal intubation. After anesthesia induction, post-induction cerebral hemodynamic and metabolic parameters will be obtained.

After tracheal intubation with airway secured, maintenance and vasopressor agents will be administrated according to the allocated group. The four possible allocated groups are as follows:

Group 1: Propofol-based anesthetic maintenance with phenylephrine used as the vasopressor Group 2: Propofol-based anesthetic maintenance with ephedrine used as the vasopressor Group 3: Sevoflurane-based anesthetic maintenance with phenylephrine used as the vasopressor Group 4: Sevoflurane-based anesthetic maintenance with ephedrine used as the vasopressor

Maintenance agents

* For the propofol group, the patient will receive propofol as their maintenance agent during surgery. The typical dose is 150-200 mg/kg/min.
* For the sevoflurane group, the patient will be maintained with 1 MAC of sevoflurane during surgery.
* Both propofol and sevoflurane are commonly used maintenance agents, and the depth of anesthesia will be kept at PSI of 30-40 (normal range 25-50) regardless of the choice of agents. Anesthesiologists use both agents frequently, and in our daily practice, the choice of anesthetic agents is mainly based on personal preference, with the exception of patients with specific contraindications such as malignant hyperthermia or drug allergy.

Vasopressor agents

* For the phenylephrine group, the patient will receive phenylephrine infusion as the primary vasopressor of choice.
* For the ephedrine group, the patient will receive ephedrine infusion as the primary vasopressor of choice.
* Vasopressor will only be administrated to maintain MAP within 0-20% above the baseline. In general anesthesia practice, ephedrine and phenylephrine can be administrated as a bolus injection or infusion. In this study, an infusion regime is used because of the necessity of maintaining a stable blood pressure during repeated measurements of cerebral hemodynamics in a steady state in each group. In patients with refractory hypotension despite either phenylephrine or ephedrine infusion, other vasopressor or inotropes will be used. For patients who did not receive any vasopressor (e.g. no hypotension during the entire surgery) or who receive multiple types of vasopressors, the investigators will analyze their data using both an intention-to-treat and as-per-protocol approach.

The neurological outcomes of patients in the post-anesthesia care unit (PACU) will also be collected via routine physical exam.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients over the age of 18 years old.
2. ASA I-IV
3. Undergoing surgery under general anesthesia at London Health Sciences Centre or St. Joseph's Healthcare that is scheduled to last longer than 1 hour.

Exclusion Criteria:

1. Had any neurological conditions such as history of stroke, TIA, neurodegenerative disease, or carotid stenosis
2. Had a history of substance abuse such as heavy cannabis users
3. Have a contraindication of applying the cerebral oximetry device (e.g., skin lesions in the forehead)
4. Have contraindications to receive specific anesthetic agents or vasopressors such as malignant hyperthermia or an allergy.
5. Unable to communicate with the research staff

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Effects of anesthetic maintenance agents and vasopressors on cerebral hemodynamics and metabolism. | Duration of surgery
  Differences in CMRO2 during surgery between sevoflurane and propofol groups will be analyzed by repeated measures ANOVA. Next, differences in CMRO2 during surgery between the phenylephrine and ephedrine groups will be compared by repeated measures ANOVA. To explore any interaction, we will examine whether the effect of one independent variable depends on the level of the other independent variable by conducting a two-way ANOVA. A two-way ANOVA will allow us to examine the main effects of each independent variable and the interaction effect. The interaction effect can be examined by looking at the F-value and p-value associated with the interaction term in the ANOVA output. If the p-value is significant (i.e., less than the alpha level), then there is evidence of an interaction effect.

SECONDARY OUTCOMES:
Effects of anesthetic maintenance agents and vasopressors on cerebral hemodynamics and metabolism during induction | Anesthesia induction
  The times corresponding to the anesthesia induction with propofol will be marked. Short periods (60 s before and 300 s after propofol injection) are selected to measure CBF and CMRO2 changes. The onset of anesthesia will be confirmed with BIS/PSI monitor. To test the hypotheses, one-way repeated measures ANOVA will be used to compare the differences between before and after anesthesia induction. The time sequence of cerebral hemodynamics and metabolism in relation to the changes of systemic blood pressure will be plotted out. In addition, multiple regression analysis will be used to investigate the relationship between patient characteristics (baseline arterial blood pressure, medical comorbidities) and the magnitude of CBF and CMRO2 reductions during anesthesia induction.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Chui, MD, Principal Investigator — Western University
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.

REFERENCES:
- [Background] Murkin JM. Cerebral oximetry: monitoring the brain as the index organ. Anesthesiology. 2011 Jan;114(1):12-3. doi: 10.1097/ALN.0b013e3181fef5d2. No abstract available. PMID 21178667
- [Background] Jonsson M, Lindstrom D, Wanhainen A, Djavani Gidlund K, Gillgren P. Near Infrared Spectroscopy as a Predictor for Shunt Requirement During Carotid Endarterectomy. Eur J Vasc Endovasc Surg. 2017 Jun;53(6):783-791. doi: 10.1016/j.ejvs.2017.02.033. Epub 2017 Apr 19. PMID 28431821
- [Background] Khozhenko A, Lamperti M, Terracina S, Bilotta F. Can Cerebral Near-infrared Spectroscopy Predict Cerebral Ischemic Events in Neurosurgical Patients? A Narrative Review of the Literature. J Neurosurg Anesthesiol. 2019 Oct;31(4):378-384. doi: 10.1097/ANA.0000000000000522. PMID 30001276
- [Background] Khan JM, McInnis CL, Ross-White A, Day AG, Norman PA, Boyd JG. Overview and Diagnostic Accuracy of Near Infrared Spectroscopy in Carotid Endarterectomy: A Systematic Review and Meta-analysis. Eur J Vasc Endovasc Surg. 2021 Nov;62(5):695-704. doi: 10.1016/j.ejvs.2021.08.022. Epub 2021 Oct 6. PMID 34627675
- [Background] Milej D, Shahid M, Abdalmalak A, Rajaram A, Diop M, St Lawrence K. Characterizing dynamic cerebral vascular reactivity using a hybrid system combining time-resolved near-infrared and diffuse correlation spectroscopy. Biomed Opt Express. 2020 Jul 23;11(8):4571-4585. doi: 10.1364/BOE.392113. eCollection 2020 Aug 1. PMID 32923065
- [Background] Milej D, He L, Abdalmalak A, Baker WB, Anazodo UC, Diop M, Dolui S, Kavuri VC, Pavlosky W, Wang L, Balu R, Detre JA, Amendolia O, Quattrone F, Kofke WA, Yodh AG, St Lawrence K. Quantification of cerebral blood flow in adults by contrast-enhanced near-infrared spectroscopy: Validation against MRI. J Cereb Blood Flow Metab. 2020 Aug;40(8):1672-1684. doi: 10.1177/0271678X19872564. Epub 2019 Sep 9. PMID 31500522
- [Background] Abdalmalak A, Milej D, Diop M, Shokouhi M, Naci L, Owen AM, St Lawrence K. Can time-resolved NIRS provide the sensitivity to detect brain activity during motor imagery consistently? Biomed Opt Express. 2017 Mar 13;8(4):2162-2172. doi: 10.1364/BOE.8.002162. eCollection 2017 Apr 1. PMID 28736662
- [Background] Durduran T, Yodh AG. Diffuse correlation spectroscopy for non-invasive, micro-vascular cerebral blood flow measurement. Neuroimage. 2014 Jan 15;85 Pt 1(0 1):51-63. doi: 10.1016/j.neuroimage.2013.06.017. Epub 2013 Jun 14. PMID 23770408
- [Background] Selb J, Boas DA, Chan ST, Evans KC, Buckley EM, Carp SA. Sensitivity of near-infrared spectroscopy and diffuse correlation spectroscopy to brain hemodynamics: simulations and experimental findings during hypercapnia. Neurophotonics. 2014 Jul;1(1):015005. doi: 10.1117/1.NPh.1.1.015005. PMID 25453036
- [Background] Verdecchia K, Diop M, Lee A, Morrison LB, Lee TY, St Lawrence K. Assessment of a multi-layered diffuse correlation spectroscopy method for monitoring cerebral blood flow in adults. Biomed Opt Express. 2016 Aug 24;7(9):3659-3674. doi: 10.1364/BOE.7.003659. eCollection 2016 Sep 1. PMID 27699127
- [Background] Rajaram A, Milej D, Suwalski M, Kebaya L, Kewin M, Yip L, de Ribaupierre S, Han V, Diop M, Bhattacharya S, St Lawrence K. Assessing cerebral blood flow, oxygenation and cytochrome c oxidase stability in preterm infants during the first 3 days after birth. Sci Rep. 2022 Jan 7;12(1):181. doi: 10.1038/s41598-021-03830-7. PMID 34996949
- [Background] Rajaram A, Milej D, Suwalski M, Yip LCM, Guo LR, Chu MWA, Chui J, Diop M, Murkin JM, St Lawrence K. Optical monitoring of cerebral perfusion and metabolism in adults during cardiac surgery with cardiopulmonary bypass. Biomed Opt Express. 2020 Sep 29;11(10):5967-5981. doi: 10.1364/BOE.404101. eCollection 2020 Oct 1. PMID 33149999
- [Background] Kaya K, Zavriyev AI, Orihuela-Espina F, Simon MV, LaMuraglia GM, Pierce ET, Franceschini MA, Sunwoo J. Intraoperative Cerebral Hemodynamic Monitoring during Carotid Endarterectomy via Diffuse Correlation Spectroscopy and Near-Infrared Spectroscopy. Brain Sci. 2022 Aug 2;12(8):1025. doi: 10.3390/brainsci12081025. PMID 36009088